CLINICAL TRIAL: NCT02024230
Title: Rivaroxaban Estimation With Warfarin in Atrial Fibrillation Patients With Coronary Stent Implantation Study (REWRAPS)
Acronym: REWRAPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fujita Health University (Other)
Responsible Party: Principal Investigator, Yukio Ozaki, Department of Cardiology, Fujita Health University, Fujita Health University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REWRAPS
Record Dates: First submitted 2013-12-10; First posted 2013-12-31 (Estimated); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation; Stroke; Fetal Blood Loss; Major Bleeding; All Cause Mortality
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation; Stroke | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Active Comparator): Patients were treated over a median of 4.75 years with either rivaroxaban (10 mg once daily for patients with a creatinine clearance of 15-49 mL/min or 15 mg once daily for patients with a creatinine clearance ≥50 mL/min)
  Interventions: Drug: Rivaroxaban or Warfarin
- Warfarin (Active Comparator): The dose of warfarin can be controlled with dose adjustment to achieve a target international normalized ratio [INR] of 2.0-3.0 or in patients aged >70 years and having a high bleeding risk, a target INR of 1.6-2.6) according to the guideline of Japanese Circulation Society based on the following paper (Inoue H, Okumura K, Atarashi H, Yamashita T, Origasa H, Kumagai N, et al. Target international normalized ratio values for preventing thromboembolic and hemorrhagic events in Japanese patients with non-valvular atrial fibrillation: results of the J-RHYTHM Registry. Circ J 2013;77(9):2264-70.)
  Interventions: Drug: Rivaroxaban or Warfarin

INTERVENTIONS:
Drug: Rivaroxaban or Warfarin — a multi-center, prospective, non-randomized, open-label, physician-initiated interventional allocation study either rivaroxaban or warfarin

SUMMARY:
Antiplatelet therapy is indispensable for the prevention of stent thrombosis in patients who underwent coronary artery stenting. Similarly, anticoagulant therapy is essential for the prevention of cardiogenic embolism including cerebral infarction in AF patients. However, the combined antithrombotic therapy has been reported to increase the risk of major bleeding for AF patients after coronary stenting, New anticoagulant drugs that hardly interact with other drugs and do not need frequent blood tests have become commonly used. The purpose of this study is to assess the hypothesis that Rivaroxaban is non-inferior to Warfarin in the efficacy and safety for AF patients after coronary stenting

ELIGIBILITY:
Inclusion Criteria:

Clinically stable atrial fibrillation (AF) patients who underwent coronary artery stenting more than one year ago and are treated or are scheduled to be treated with anticoagulant drug (regardless of the type of stents and AF).

Those who are willing to cooperate with us in the study. Those who can sign the informed consent document that is approved by the ethics committee of the medical institution participating in the study.

Exclusion Criteria:

Those in whom the package inserts state anticoagulant drugs are contraindicated for use Those who are scheduled to undergo percutaneous coronary intervention or catheter ablation for AF. Those who have to continuously undergo dual antiplatelet due to a past history of stent thrombosis during the distant stage after stenting. Those who have undergone prosthetic valve replacement for valvular disease. Those who the physician in charge judges are ineligible for the study due to serious pathological conditions. Those who are not willing to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
a composite of adverse events | 3 years
  cardiac or stroke death, non-fatal myocardial infarction, non-fatal stroke, coronary artery revascularization (percutaneous coronary intervention or coronary artery bypass graft), and systemic embolism
major bleeding | 3 years
  BARC 3 and 5
Net Adverse Clinical Event (NACE) | 3 years
  a composite of all-cause death and major bleeding

SECONDARY OUTCOMES:
all-cause death | 3 years
admission due to congestive heart failure | 3 years
fatal arrhythmia | 3 years
electrocardiographic findings | 3 years
  rhythm, ST change, Q wave abnormality, QRS duration, QT interval, QTc interval, the presence of supraventricular premature contraction (SVPC), the presence of ventricular premature contraction (VPC)
cardiac ultrasound findings | 3 years
  left atrial dilatation (LAD), left ventricular end-diastolic diameter (LVDd), left ventricular end-systolic diameter (LVDs), E/A, E/E', tricuspid regurgitation pressure gradient (TRPG), LV wall abnormality
each cardiovascular event used for the primary efficacy outcome measures | 3 years
non-major clinical relevant bleeding | 3 years
cardiac or stroke death | 3 years
non-fatal myocardial infarction | 3 years
non-fatal stroke | 3 years
coronary artery revascularization (percutaneous coronary intervention or coronary artery bypass graft) | 3 years
systemic embolism | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Yukio Ozaki, Nagoya, Aichi-ken, Japan